CLINICAL TRIAL: NCT01301417
Title: a RETROspective Data Collection of comPRESSion Anastomosis Using the ColonRing ™
Brief Title: Data Collection of Patients Treated With the ColonRing™ for the Creation of Circular Compression Anastomosis
Acronym: RETROPRESS
Status: Completed | Type: Observational
Sponsor: novoGI (Industry)
Responsible Party: Sponsor
Other Study IDs: RETROPRESS
Record Dates: First submitted 2011-02-20; First posted 2011-02-23 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Diverticulum, Colon; Colorectal Neoplasms; Crohn Disease; Colitis, Ulcerative; Colostomy; Ileostomy - Stoma; Rectal Prolapse; Intestinal Polyposis; Lymphoma; Endometriosis; Intestinal Volvulus
Keywords: Compression Anastomosis
MeSH Terms: conditions — Diverticulum, Colon; Colorectal Neoplasms; Crohn Disease; Colitis, Ulcerative; Rectal Prolapse; Intestinal Polyposis; Lymphoma; Endometriosis; Intestinal Volvulus

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ColonRing™: Adult Patients who underwent a laparoscopic or open colorectal resection with the creation of an anastomosis using the ColonRing™ in routine clinical practice
  Interventions: Device: ColonRing™

INTERVENTIONS:
Device: ColonRing™ — Creation of a circular Compression Anastomosis
  Other Names: Compression Anaqstomosis Ring™(CAR™)27

SUMMARY:
The proposed study is a post marketing, observational, retrospective data collection intended to gather and record data on patients treated with the ColonRing™ device in routine clinical practice at a single center. The data will assist in further evaluating the performance of the ColonRing™ device in regards to the creation of a colorectal anastomosis.

Hypothesis:The performance of the ColonRing™, determined by the rate of complications, will be within the acceptable range reported in the literature for alternative treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Patient was > 18 years old at time of procedure
* Patient underwent an open or laparoscopic colorectal procedure with the creation of an anastomosis using the ColonRing™
* Patient treated in routine clinical practice following marketing clearance of the device within the cleared intended use
* Patient underwent his/her first follow-up visit within two months post-surgery

Exclusion Criteria:

* No exclusion criteria have been defined for this data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients who underwent a laparoscopic or open colorectal resection with the creation of an anastomosis using the ColonRing™ in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Rate of anastomotic leakage | 2-mo post-op
  The primary study outcome is the rate of anastomotic leakage. Anastomotic leakage is defined as evidence of a defect in the intestinal wall integrity at the anastomotic site leading to a communication between the intra and extra luminal compartments.

SECONDARY OUTCOMES:
Rate of other device related complications and measures during hospitalization and post procedure: | 2-mo post-op
  The following complications will be examined for relation to the device:
  Bleeding. Stricture (either clinical evidence of a stricture or the inability to pass a 12 mm sigmoidoscope through the anastomosis in a procedure that does not include a diversion). Septic complication (including wound infection, pelvic infection, peritonitis, abscess).
  Readmission, re-operation, death within two months of the procedure. Extra colonic complications (including urinary infection, urinary retention, DVT, pneumonitis, pulmonary embolism, cardiac, injury to other organs - e.g. spleen, ureter)

CONTACTS AND LOCATIONS:
Overall Officials: Eran Choman, Msc, Study Director — novoGI
Locations (1):
- Southern Regional Medical Center, Riverdale, Georgia, United States